CLINICAL TRIAL: NCT01854021
Title: Effects of Different General Anesthesia Methods on Immune Responses in Patients Undergoing Surgery for Tongue Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: tiejun Zhang (Other)
Responsible Party: Sponsor-Investigator, tiejun Zhang, Department of Anesthesiology , School and Hospital of Stomatology, Wuhan University, Wuhan University
Organization: Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: wuhan university
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Tongue Cancer
Keywords: Anesthesia; general; Immunity; Tongue neoplasms; immune; general anesthesia
MeSH Terms: conditions — Tongue Neoplasms | interventions — Anesthesia, Intravenous

ARMS (3):
- inhalational anesthesia (Experimental): inhalational anesthesia
  Interventions: Procedure: inhalational anesthesia
- combined intravenous-inhalational anesthesia (Experimental): combined intravenous-inhalational anesthesia
  Interventions: Procedure: combined intravenous-inhalational anesthesia
- intravenous anesthesia (Experimental): intravenous anesthesia
  Interventions: Procedure: intravenous anesthesia

INTERVENTIONS:
Procedure: intravenous anesthesia — intravenous anesthesia
  Arms: intravenous anesthesia
Procedure: combined intravenous-inhalational anesthesia — combined intravenous-inhalational anesthesia
  Arms: combined intravenous-inhalational anesthesia
Procedure: inhalational anesthesia — inhalational anesthesia
  Arms: inhalational anesthesia

SUMMARY:
Surgical excision is the mainstay of treatment for tongue cancer. However, surgery-induced immunosuppression has been implicated in the development of post-operative septic complications and neoplasm metastasis. General anesthesia is considered to not only suppress surgical stress, but also affect the immune function directly，such as altering the number and activity of immune cells. It is reported that some anesthetics increase susceptibility to tumor metastasis, apparently by suppressing natural killer cell activity. Different anesthetic techniques and anesthetics used in anesthesia have shown different effects on immunity. Many of the studies were animal trials or performed in vitro; in addition, most are focused on a single drug. To date, there is little published prospective clinical research designed specifically to investigate the effects of different general anesthetic technique on immune function in patients with oral malignant tumors. The aim of this study is going to characterize the immune response of patients undergoing surgery for tongue cancer under 3 types of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All the patients were scheduled for elective surgery for tongue cancer under general anesthesia. None of the patients had a history of endocrine, immune and circulatory system diseases;
* Exclusion criteria were also contraindications for receiving chemotherapy

Exclusion Criteria:

* contraindications for receiving chemotherapy,
* receiving perioperative blood transfusion, or
* preoperative and perioperative treatment with hormones and immunomodulatory agent.

Patients who suffered from any surgical complications such as infection were also excluded from our study.

-

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Percentages of immune cells | 3 days
  30 min before induction, 1 h, 3 h and 5 h after induction; at the end of operation and 24h, 48 h and 72 h after operation

SECONDARY OUTCOMES:
Percentages of T lymphocytes subsets | 3 days
  30 min before induction, 1 h, 3 h and 5 h after induction; at the end of operation and 24h, 48 h and 72 h after operation
Percentages of Natural Killer cells | 3 days
  30 min before induction, 1 h, 3 h and 5 h after induction; at the end of operation and 24h, 48 h and 72 h after operation
Percentages of B lymphocytes | 3 days
  30 min before induction, 1 h, 3 h and 5 h after induction; at the end of operation and 24h, 48 h and 72 h after operation

CONTACTS AND LOCATIONS:
Overall Officials: kebin Liu, Study Director — Master of Department of Anesthesiology of Hospital of Stomatology, Wuhan University
Locations (1):
- Hospital of stomatology of wuhan university, Wuhan, Hubei, China